Protocol Title: GPR109A and Parkinson's Disease: Role of Niacin in Outcome

Measures

Principal Investigator: Chandramohan Wakade

## 1. Objectives

Describe the purpose, specific aims, and hypothesis:

(1) examine the blood, urine and spinal fluid of persons with Parkinson's to look for evidence of inflammation and; (2) whether 6 months of vitamin B3 supplementation may reduce the inflammation and/or improve symptoms.

## 2. Background

Describe the background and rationale for the study:

Inflammation plays a central role in Parkinson's disease (PD) pathology [1] as evidenced by the presence of microglia in the substantia nigra in post-mortem samples [2] as well as activated microglia and cytokines in clinical and animal studies [3]. The use of non-aspirin non-steroidal anti-inflammatory drugs was found to reduce the risk of PD [4]. We recently identified an anti-inflammatory receptor GPR109A that is upregulated in PD [5]. Niacin has a high affinity for this receptor, suggesting that it (niacin) may play an important role in reducing inflammation in PD. We also found that individuals with PD have a chronic niacin deficiency [5]. Using seed funding from the local PD chapter, we obtained pilot data which suggested that restoring the deficiency via over-the-counter (OTC) supplementation reduced inflammation and decreased the severity of the disease symptoms [6]. In this VA-funded study, we will determine the effect of 6 months' OTC niacin supplementation on inflammation (as assessed in the blood and spinal fluid) and severity of the PD symptoms.

#### References

- 1. Barnum CJ, Tansey MG (2010) Modeling neuroinflammatory pathogenesis of Parkinson's disease. Prog Brain Res 184: 113–132
- 2. Banati RB, Daniel SE, Blunt SB (1998) Glial pathology but absence of apoptotic nigral neurons in long-standing Parkinson's disease. Movement Disorders 13: 221–227.
- 3. Crotty S, Fitzgerald P, Tuohy E, Harris DM, Fisher A, et al. (2008). Neuroprotective effects of novel phosphatidylglycerol-based phospholipids in the 6-hydroxydopamine model of Parkinson's disease. European Journal of Neuroscience 27: 294–300.
- 4. Gagne JJ, Powers MC (2010) Anti-inflammatory drugs and risk of Parkinson's disease: A meta-analysis Neurol 74: 995–1002.
- 5. Wakade, C., Chong, R. K., Thomas, B., Bradley, E., & Morgan, J. (2014). Upregulation of GPR109A in Parkinson's disease. PloS ONE, 9(10), e109818.
- 6. Wakade, C., Chong, R. K., Bradley, E., & Morgan, J. (2015). Low-dose niacin supplementation modulates GPR109A levels and NAD/NADH ratio and ameliorates PD symptoms. Clinical Case Reports. doi: 10.1002/ccr1003.1232.

 Version Date: 1/13/16; 6/24/16

### 3. Inclusion and Exclusion Criteria

List the inclusion/exclusion criteria:

Inclusion criteria

PD subjects will be adult men and women diagnosed with idiopathic mild to moderately severe PD defined as modified Hoehn & Yahr Stages I-III (while "On"). PD is defined according to the UK Brain Bank Criteria made at least six months prior to recruitment to the study. PD features include the presence of at least two of the four cardinal clinical manifestations of the disease, which are tremor, rigidity, bradykinesia, and disturbances of posture or gait, without any other known or suspected cause of Parkinsonism. Subjects should be stabilized on PD medication for at least 3 months before enrollment into the study. Subjects' PD drug prescriptions will not be altered nor withheld during the study, i.e., they will be tested while "On." The patient will have signed informed consent. Subjects who do not have PD (i.e., healthy or have other medical conditions such as TBI, stroke, or other syndromes in which inflammation plays a role in the condition will also be recruited as control subjects. This will allow us to estimate whether these other conditions show similar or unique inflammatory profile.

#### Exclusion criteria

Subjects will be excluded if they had previous brain surgery or other severe neurological problems – intracerebral hemorrhage, traumatic brain injury, central nervous system malignancy, active CNS infection, significant stroke, Alzheimer disease or any type of implanted stimulator including but not limited to Deep Brain Stimulator (DBS) or pacemaker. All subjects must be without evidence of dementia, defined as a score > 24 the Mini-Mental State Examination and able to understand test instructions. Subjects must not have functional blindness (inability to participate in gait and visuomotor assessments) or lower limb amputation higher than the forefoot or any orthopedic problem that precludes performance of physical tests. Allergic to niacin. Significant cardiac, pulmonary, hepatic, gastrointestinal, or renal disease (e.g., New York Heart Association Class III or IV congestive heart failure; endocarditis; pulmonary insufficiency symptomatic at rest or with mild physical exertion; acute or chronic hepatitis; renal failure requiring dialysis; second and third degree AV block or sick sinus syndrome), or diabetes are also exclusionary factors.

# 4. Number of Subjects/Records/Samples Collected

Indicate the total number of subjects to be accrued/records reviewed/samples collected across all sites: 100

### 5. Recruitment Methods

Describe when, where, and how potential subjects will be recruited:

VA clinic (including medical records), word of mouth.

### 6. Procedures Involved

a. Describe the procedures involved to include those procedures that are standard evaluation and/or care and those that are solely for research purposes:

Standard procedures: basic physical examination for strength, speed, coordination, tremor, flexibility, rigidity and reaction time


| | Research procedures: questionnaire and tests to document health and cognitive status, blood, urine and spinal fluid samples, over-the-counter (non-prescription) vitamin B3 supplementation |
|---|---|
| b. | Describe and explain the study design: |
| | Pre-post repeated measures placebo-controlled study |
| c. | Describe the procedures performed to lessen the probability or magnitude of risks: |
| | Use of slow-release supplement to minimize potential skin itching |
| d. | Describe the duration of an individual subject's participation in the study and the time involved: |
| | 6 months supplement study with a pre and post test, each lasting about 1 to 1.5 hr. |

# 7. Data and Specimen Management

| • | Dau | and Specimen Management | |
|---|---|---|---|
| | a. | Describe the data analysis plan, including any statistical procedures: We will use the Unified Parkinson's Disease Rating Scale (UPDRS) III (Motor Section) as the primary pre- and post-treatment outcome assessment that is recommended for PD studies. Significant changes in outcome measures will be determined by performing a Mixed model analysis of variance, with Groups as the independent factor and Time as the repeated factor. | □ N/A |
| | b. | When applicable, provide a power analysis: | □ N/A |
| | | Based on the preliminary data using unpaired simple effects analyses, the minimum number of subjects needed per group to detect a statistical significance @ $p = .05$ , 2-tailed and 80% power of detection are as follows: | |
| | | Outcome measures Effect size (based on Cohen's d) # Subjects/group UPDRS motor 1.46 14 Sleep efficiency (pilot data) 0.97 8 | |
| | | The sample sizes are based on a large effect size, i.e., a grossly observable and clinically meaningful treatment effect. We have demonstrated that this is a reasonable expectation based on the actual effect sizes of the human preliminary data that we have shown. We used simple effects analyses as the basis for the sample size calculations because any sample size calculations based on the full design would require knowledge of the intraclass correlation across the treatments, as well as the carry-over, group, and period effects. | |
| | | Correlation statistics. Based on the preliminary data's correlation coefficients (r) obtained via simple linear independent correlation tests comparing the variables versus disease severity (UPDRS motor section), the minimum number of subjects needed per group to detect a statistical significance @ $p = .05$ , and 80% are as follows: | |


| | ome measures | r | # Subjects/group | |
|---|---|---|---|---|
| | 109A levels | 0.59 | 20 | |
| | Sleep Time | -0.57 | 18 | |
| | to Fall Asleep | 0.79 | 8 | |
| Sleep | Efficiency | -0.73 | 10 | |
| propo<br>poten<br>unexj<br>100 s | ose to collect 30 PD<br>tial subject dropout<br>pected increase in the<br>ubjects to take into<br>ase in the variability | subjects per grass, experimental ne variability of account potent | tion power analyses above, we roup (total 60) to account for l/data corruption and/or an f the data. We plan to recruit a ial drop-outs and an unexpectation impacts the estimated states. | about<br>ted |
| c. Descr | ribe how data and s | pecimens will l | be handled: | □ N/A |
| i. | What information | ı will be includ | ed in that data or associated | with the specimens? |
| | Please refer to 6 | a above All da | ta will be coded | |
| ii. | | | cimens will be stored? | |
| | | | cured computer. ICD will be so specimens will be coded. | stored in a locked |
| iii. | | | pecimens be stored? | |
| | Indefinitely | | | |
| iv. | Who will have ac | cess to the data | a or specimens? | |
| | | | T | |
| | Research team | | | |
| v. | Who is responsib | le for receipt o | r transmission of the data and | d/or specimens? |
| • • | | | | |
| | Chandramohan \ | (Vakade (PI) | | |
| vi. | Chandramohan \ How will data an | | s be transported? | |
| | | | s be transported? | |


| • | Prov | visions to Monitor the Data to Ensure the Safety of Subjects |
|---|---|---|
| | This | study involves no more than minimal risk study and this section is not required. $\square$ $N/A$ |
| | - | plan might include establishing a data monitoring committee and a plan for reporting data toring committee findings to the IRB and the sponsor. |
| | a. | Describe the plan to periodically evaluate the data collected regarding both harms and benefits to determine whether subjects remain safe. |
| | | Subjects will be contacted the day after their pre- and post-test participation in the study to make sure that they did not experience unexpected or severe reactions to the vitamin supplement and optional lumbar puncture. A log will be kept to document the contact and relevant information from the subject. Subjects will also be given a 24-hour hotline to report any adverse event that they think is related to the study. |
| | b. | Describe what data are reviewed, including safety data, untoward events, and efficacy data. |
| | | fety and untoward events related to the vitamin supplement and optional lumbar puncture ll be reviewed. |
| | С. | Describe how the safety information will be collected (e.g., with case report forms, at study visits, by telephone calls with participants). |
| | | Safety information will be collected by telephone calls or emails with the participants. |
| | d. | Describe the frequency of data collection, including when safety data collection starts. |
| | | Data will be collected by the researchers at baseline and the end of the study. Subjects will be instructed to contact the researchers as soon as possible if they experience any adverse events that they think is related to the study. |
| | e. | Describe who will review the data. |
| | | Dr Chandramohan Wakade will be the main person to review the data. He will consult with Dr John Morgan or Dr Raymond Chong if needed. |
| | f. | Describe the frequency or periodicity of review of cumulative data. |
| | | Cumulative data will be reviewed every month to ensure adherence to the approved protocol. |
| | g. | Describe any conditions that trigger an immediate suspension of the research. |
| | | If a subject reports an unexpected adverse event, the study will be suspended. The study will resume if it is determined that the event is unrelated to the study. |


| . Wit | hdrawal of Subjects | / <b>A</b> |
|---|---|---|
| a. | If applicable, describe anticipated circumstances under which subjects will be withdrawn from the research without their consent. Click here to enter text. | ⊠ N/A |
| b. | If applicable, describe any procedures for orderly termination. | ⊠ N/A |
| | Click here to enter text. | |
| c. | If applicable, describe procedures that will be followed when subjects withdraw from the research, including partial withdrawal from procedures with continued data collection. | □ N/A |
| | A subject who withdraws from the study on their own accord will be replaced by another. A subject who partially withdraws from procedures will remain in the study as long as they continue taking the supplement. | |
| 0. Ris | sks to Subjects | |
| Low-l<br>lumba<br>will be<br>Thron<br>spinal<br>Discor<br>blood<br>leakag<br>We we<br>Overa<br>his op | a. List the reasonably foreseeable risks. ow-level temporary discomfort or pain during the blood and lumbar draw. Contraindications for the ambar puncture: Although there are no absolute contraindications to performing the procedure, caution will be used in patients with the following conditions: 1) Possible raised intracranial pressure; 2) Phrombocytopenia or other bleeding diathesis (including ongoing anticoagulant therapy); 3) Suspected pinal epidural abscess. The side effects associated with lumbar puncture may include following: 1) Discomfort or pain during the procedure; 2) Bleeding into the spinal cord, particularly in people who take lood thinners or have a low platelet count (thrombocytopenia); 3) Temporary headache as a result of CSF cakage; 4) Infection; 5) Nerve damage; 6) Cerebral herniation; 7) Temporary back pain. We will take a conservative approach in deciding which patient to include from the lumbar procedure. Overall, Dr. John Morgan will exercise his clinical judgment to exclude a subject from the procedure if, in is opinion, he feels that the subject presents with a set of conditions which renders them unsuitable for the rocedure. | |
| b. | If applicable, describe any costs that subjects may be responsible for because of participation in the research. | ⊠ N/A |
| | Click here to enter text. | |
| С. | If applicable, describe risks to others who are not subjects. | □ N/A |
| | Click here to enter text. | |


## 11. Potential Benefits to Subjects

Describe the potential benefits that individual subjects may experience from taking part in the research. Niacin is an over-the-counter supplement. Our preliminary data indicates that PD patients will benefit from the supplementation. The dosage selected is 250 mg daily dose for 6 months. These dosages are low and do not produce any side effects. If at all, the PD patients will be benefitted by its actions. Subjects will be given a \$50 gift card for successfully completing the 6-month study. They will receive an additional \$100 if they participate in the spinal draw. At the end of the study, all subjects will receive the real niacin and be invited back for an optional follow-up assessment.

## 12. Confidentiality

Describe the procedures for maintenance of confidentiality.

All data will be kept in locked files and information on computer databases including cloud storage will be coded to protect patient identity. The only place where the subject's identity is revealed is the Informed Consent form. Subjects' identity will be coded in all other sources of documentation (hard copies and electronic files).

### 13. Consent Process

*If you are obtaining consent of subjects describe the consenting process.* 

Subjects who indicate an interest to participate in this study will be tested at the VA clinic and/or visit Dr. Raymond Chong's ground-floor Human Movement Science lab on the GRU campus. Blood and urine samples will be obtained in the adjacent room in the Interdisciplinary Clinical Practice facility. The nature of the information in the informed consent will be a brief overview of the study, tests involved, benefit and risks as well as the subject's right to terminate the session at any time. The informed consent will also state that each participant agrees to freely and voluntarily participate in the study. The document will also state that any other financial impact is the participant's sole responsibility.

# 14. Compensation for Research-Related Injury

This section is not required when research involves no more than Minimal Risk to subjects.  $\boxtimes N/A$ 

a. Describe the available compensation in the event of research related injury.

Click here to enter text.

#### 15. Resources Available

 $\bowtie$  N/A

- a. Describe the availability of medical or psychological resources that subjects might need as a result of an anticipated consequences of the human research.

  Click here to enter text.
- b. Describe your process to ensure that all persons assisting with the research are adequately informed about the protocol, the research procedures, and their duties and functions.

Documentation from the VA facility will be provided that research team members have undergone training in the following areas: Good clinical Practices; the ethical principles of


human research protection; Privacy; Cybersecurity; and VA Research Data Security and Privacy.
